CLINICAL TRIAL: NCT03387462
Title: DOT Diary (D2): Developing a Mobile App With Combined Automated DOT and Daily Sexual Diary for Monitoring and Improving PrEP Adherence: DOT Diary Optimization Pilot
Brief Title: DOT Diary Optimization Pilot: A Pilot Study to Optimize the DOT Diary App to Measure PrEP Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); San Francisco Department of Public Health (Other Government); Emory University (Other); AiCure (Industry)
Responsible Party: Principal Investigator, Susan Buchbinder, Director, Bridge HIV, Public Health Foundation Enterprises, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-22864; 1R01MH109320-01 (NIH)
Record Dates: First submitted 2017-12-01; First posted 2018-01-02 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Adherence, Medication; Risk Behavior; Pre-Exposure Prophylaxis; HIV Prevention
Keywords: Adherence; PrEP; HIV Prevention; Truvada; HIV Risk Reduction; Mobile App
MeSH Terms: conditions — Medication Adherence; Risk-Taking | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DOT Diary Optimization Intervention (Experimental): DOT Diary mobile app and Emtricitabine / Tenofovir Disoproxil Oral Tablet
  Interventions: Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet; Other: DOT Diary mobile app

INTERVENTIONS:
Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet — Open label daily emtricitabine/tenofovir disoproxil oral tablet
  Other Names: Truvada
Other: DOT Diary mobile app — DOT Diary mobile application for tracking medication adherence and sexual activities.

SUMMARY:
The researchers are working with a technology company, AiCure, to develop a smartphone app, DOT Diary, which combines two drug adherence strategies. DOT Diary reminds people when it is time to take their medication, and uses motion-sensing technology to visually and automatically confirm the pill was swallowed. The goal of this study is to understand people's experiences using this new app while taking HIV pre-exposure prophylaxis (PrEP) for the prevention of HIV.

DETAILED DESCRIPTION:
In the DOT Diary research project, the AiCure aDOT smartphone app has been adapted for use in monitoring and supporting HIV pre-exposure prophylaxis (PrEP) use among young men who have sex with men (YMSM). The aDOT app uses automated directly observed therapy (DOT) that use the smartphone camera and artificial intelligence software to confirm that the right person is taking the right medication at the right time. A sexual diary has been integrated into the aDOT app to assist YMSM in understanding whether they are receiving protection from PrEP for individual sexual episodes, and when it is particularly important to take PrEP (e.g. after a sexual episode).

In the next stage of app development, the researchers are conducting this study to identify areas of the app that require refinement to maximize the acceptability and ease of use of the DOT adherence monitoring app. The researchers will assess overall acceptability and ease of use of the integrated DOT Diary (D2) app over an 8 week period.The goal of this pilot study will be to refine and optimize the app for further testing in a larger and longer pilot study among YMSM at risk for HIV acquisition. The researchers will conduct this pilot protocol among YMSM in Atlanta and San Francisco Bay Area, two metropolitan regions heavily impacted by HIV, yet differing in sociodemographics, as well as in the availability and uptake of HIV prevention services, including PrEP. These diverse research locations will allow collection of data to inform app development among a broad group of YMSM.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a man
* Age 18-35 at enrollment
* Reports having anal sex with a man or trans woman in the past 12 months and one or more of the following criteria in the past 12 months:

  * Any condomless anal sex (not in a mutually monogamous relationship with an HIV-negative partner)
  * Two or more anal sex partners
  * Self-reported STI (gonorrhea, chlamydia, syphilis)
  * Having a known HIV-positive sexual partner
* HIV-negative as determined by a negative 4th generation HIV test at screening and negative rapid 4th generation test at enrollment
* Currently taking PrEP or interested in initiating PrEP
* Eligible to take PrEP

  * Creatinine clearance ≥60 ml/min as estimated by Cockcroft-Gault equation at screening
  * Hepatitis B surface antigen (HBsAg) negative
* Willing and able to provide written informed consent
* Able to read and speak English
* Smartphone ownership compatible with DOT Diary
* Meets local locator requirements

Exclusion Criteria:

* Any reactive HIV test at screening or enrollment
* Signs or symptoms of acute HIV infection at screening or enrollment
* History of pathological bone fracture not related to trauma
* Taking nephrotoxic medications
* History of participation in the active arm of an HIV vaccine trial
* In a mutually monogamous sexual relationship with an HIV-negative partner for the past 12 months
* Does not live, work or play in Atlanta Metropolitan Area, San Francisco, Alameda, Marin, Contra Costa, Santa Clara, or San Mateo Counties
* Unable to commit to study participation for 8 weeks
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identify as a man
Enrollment: 20 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Buchbinder, MD, Principal Investigator — Bridge HIV, San Francisco Department of Public Health
Locations (2):
- United States (2):
  - Bridge HIV, San Francisco Department of Public Health, San Francisco, California
  - Emory University, School of Public Health, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
If requested, will share summary participant data with all identifying information removed.
Supporting Information: Study Protocol, ICF
Time Frame: Data are available from publication of the primary results through 3 years.
Access Criteria: Must have IRB approval.

REFERENCES:
- [Result] Liu AY, Laborde ND, Coleman K, Vittinghoff E, Gonzalez R, Wilde G, Thorne AL, Ikeguchi E, Shafner L, Sunshine L, van der Straten A, Siegler AJ, Buchbinder S. DOT Diary: Developing a Novel Mobile App Using Artificial Intelligence and an Electronic Sexual Diary to Measure and Support PrEP Adherence Among Young Men Who Have Sex with Men. AIDS Behav. 2021 Apr;25(4):1001-1012. doi: 10.1007/s10461-020-03054-2. Epub 2020 Oct 12. PMID 33044687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited online and via social media, as well as through in-person community outreach.
Period: Overall Study
Arm/Group | DOT Diary Optimization Intervention
Started | 20
4 Weeks | 20
8 Weeks | 19
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 18-35 years old, eligible, and willing to take PrEP
Arm/Group | DOT Diary Optimization Intervention
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 0
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: DOT Diary Mobile App Acceptability
Description: System Usability Scale (SUS) is a 10 item questionnaire with 5 response options: strongly disagree to strongly agree. These are scored 0-4. The scores are then summed up (making sure all positive responses -- increased usability -- are given the higher scores). The final score is multiplied by 2.5 Possible scores are from 0-100, with maximal usability achieving the higher score. Although the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
Time Frame: 8 weeks
Population: MSM eligible for or taking PrEP
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | DOT Diary Optimization Intervention
Number analyzed (Participants) | 19
Score on scale | 79.8 (15.0)

2. Primary Outcome: DOT Diary Mobile App Ease of Use
Description: 5-point Likert scale (1=strongly disagree that app is easy to use; 5=strongly agree that app is easy to use) on a single question of the key attribute of ease of use of DOT Diary over 8 weeks by MSM on PrEP.
Time Frame: 8 weeks
Population: Participants answering the ease of use question at 8 weeks.
Measure: Median (Inter-Quartile Range); unit: Score on a scale (Likert)
Arm/Group | DOT Diary Optimization Intervention
Number analyzed (Participants) | 19
Score on a scale (Likert) | 4 [4 to 5]

3. Primary Outcome: Adherence and Persistence of Use of the DOT and Sexual Diary Components of DOT Diary by Young MSM on PrEP
Description: Adherence and Persistence of use of the DOT and sexual diary components of DOT Diary by young MSM on PrEP is measured by the percentage of doses taken with visual confirmation of pill ingestion
Time Frame: 8 weeks
Population: MSM eligible for or taking PrEP
Measure: Number; unit: Percentage of doses taken
Arm/Group | DOT Diary Optimization Intervention
Number analyzed (Participants) | 19
Percentage of doses taken | 93

4. Secondary Outcome: Assessment of Situations and Reasons for Sub-optimal Use of the App
Description: Combined analysis of situations and reasons for sub-optimal use of the app, for the purpose of app optimization
Time Frame: 8 weeks
Population: MSM eligible for or taking PrEP
Measure: Number; unit: Count of participants for each reason
Arm/Group | DOT Diary Optimization Intervention
Number analyzed (Participants) | 19
Count of participants for each reason
  Technical problems | 8
  Away from home | 6

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: As daily oral FTC/TDF for PrEP is a licensed medication, the study focused assessment of AEs on the known toxicity profile of the medication, including creatinine elevations / decreases in creatinine clearance, bone fractures / toxicity, and symptoms associated with a start-up syndrome (e.g. diarrhea, nausea, headache, abdominal gas). A targeted symptom review was performed at each visit using a symptom checklist focused on symptoms associated with FTC/TDF.
Arm/Group | DOT Diary Optimization Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03387462/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT03387462/ICF_001.pdf